CLINICAL TRIAL: NCT04425369
Title: Comparison of the Inner Side and Two-sided Approaches for Iliac Crest Bone Graft Harvesting for Pediatric Pelvic Osteotomy
Brief Title: Iliac Crest Bone Graft Harvesting for Pediatric Pelvic Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuxi Su (Other)
Responsible Party: Sponsor-Investigator, Yuxi Su, Vice professor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CQMU20200017
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Child; Osteotomy
Keywords: pelvic osteotomy; developmental dysplasia of the hip; iliac crest bone graft
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inner side approaches for iliac crest bone graft (No Intervention): An anterior approach was used to expose the inner table of the ilium.
- two-sided approaches for iliac crest bone graft (Experimental): both sides of the ilium were totally exposed of the ilium.
  Interventions: Procedure: two-sided approaches for iliac crest bone graft

INTERVENTIONS:
Procedure: two-sided approaches for iliac crest bone graft — Only one side of the ilium was exposed when surgery.
  Arms: two-sided approaches for iliac crest bone graft

SUMMARY:
The iliac crest is one of the most commonly used bone graft sources, especially in pediatric pelvic osteotomy operations for developmental dysplasia of the hip (DDH) and Legg-Calve-Perthes disease. In this study, we aimed to identify the effects of inner side and two-sided approaches for iliac crest bone harvesting on post-surgery ilium growth in children.

DETAILED DESCRIPTION:
Autogenous bone grafting is still the gold standard and most effective method for treatment of non-union and bone defects due to congenital disease and infection. Despite the development of bone engineering, none of the allogeneic bone products can match the osteoinductive, osteoconductive, and immunogenic properties of autogenous bone. The iliac crest is one of the most harvested sites other than the fibula, ribs, and ulna. An iliac crest bone graft (ICBG) can supply a larger amount of cortical and cancellous bone than grafts from other donor sites. Pelvic osteotomy is widely used for treating developmental dysplasia of the hip (DDH) and Legg-Calve-Perthes disease. Tricortical structural bone such as that in the ilium is needed to stabilize the pelvis after osteotomy, and the anterior and posterior iliac crest are the two most used graft donor sites. When surgery is planned in the prone position, such as that for posterior spinal fusion, surgeons generally prefer to adopt the posterior approach for ICBG procedures. In supine position surgeries such as pelvic osteotomy for DDH or Legg-Calve-Perthes disease, surgeons prefer the anterior approach for ICBG procedures. There are many studies on iliac bone growth and complications after ICBG procedures. Most of the studies demonstrated good outcomes and few complications. However, according to our literature review, none of the previous studies used the iliac bone for transplantation in pelvic osteotomy. In this study, we compared the results between an inner table harvest site and an inner-outer table harvest site for ICBG used to maintain stability in pelvic osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* the patients who performed iliac crest bone graft and pelvic osteotomy at the same time

Exclusion Criteria:

* they had a history of pelvic osteotomy or iliac crest bone graft surgery, bilateral hip disease or congenital bone dysplasia, or were lost to follow-up.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Radiographic parameters were evaluated on anteroposterior pelvic radiographs | 3th month after surgery
  The growth areas were measured by GE healthcare-Centricity RIS CE V3.0 software (General Electric Company). The areas was calculated as mm2.
Time for the totally recovery of iliac defect | through study completion, an average of 6 months
  the time was calculated from the surgery to the time totally recovery of iliac defect by days

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No